CLINICAL TRIAL: NCT01597791
Title: Do Women Receiving Low Dose Combined Spinal Epidural for Labor Analgesia Exhibit Less Bacteriuria Using a Urinary Retention Protocol Versus Routine Urinary Catheter Placement?
Brief Title: Combined Spinal Epidural Urinary Retention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in procedure.US technically challenging.
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00005516
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2017-10-10 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia; Pain; Urinary Retention
Keywords: Urinary Retention; Urinary Catheter; Bacteriuria
MeSH Terms: conditions — Pain; Urinary Retention; Bacteriuria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foley catheter (Placebo Comparator): Control group will have a Foley catheter placed after the CSE is performed as is the usual practice at this institution.
  Interventions: Device: Foley catheter
- No Foley Catheter (Experimental): Spontaneous micturition algorithm will be assessed for spontaneous micturition and post void residual (PVR) volumes via ultrasonography at regular time intervals.
  Interventions: Other: No foley catheter

INTERVENTIONS:
Device: Foley catheter — Foley catheter placement after CSE.
  Arms: Foley catheter
Other: No foley catheter — Spontaneous Micturation/ Post Void Residual. the spontaneous micturition algorithm will be assessed for spontaneous micturition and post void residual (PVR) volumes via ultrasonography at regular time intervals.
  Arms: No Foley Catheter

SUMMARY:
The investigators hypothesize that many parturients can, in fact, spontaneously micturate with low dose combined spinal epidural analgesic doses given for labor and that Foley catheterization is unnecessary in the majority of these parturients. At Prentice Women's Hospital, almost 9000 women annually receive neuraxial labor analgesia and 98% of those receive Foley catheters. By potentially reducing the necessity for Foley catheters, the investigators should be able to ultimately reduce the rate of bacteriuria, urinary tract infections and urethritis leading to unnecessary treatment with antibiotics, as well as reduce costs of placing unnecessary Foley catheter.The hypothesis is parturients receiving low dose combined spinal epidural analgesia for analgesia after induction of labor who are randomized to a spontaneous micturition protocol will require fewer Foley catheter placements and demonstrate a lower incidence of positive urine culture postpartum than those who undergo standard Foley catheter placement.

DETAILED DESCRIPTION:
Participation in the study will begin at the patient's request for labor analgesia. The patient will be asked to urinate and a post void residual (PVR) will be measured via ultrasonography. If the PVR is >100mL, the patient will be excluded from the study. If CSF is not obtained during CSE placement or the CSE technique is abandoned for any other reason, the patient will be excluded. If the PVR is < 100mL and the combined spinal epidural analgesia is successful, they will be randomized to receive either routine Foley catheter placement or begin the spontaneous micturition protocol. Last cervical exam and VRS pain will be recorded at this time.

Subjects will be prepared in the usual fashion for the combined spinal epidural with hemodynamic monitoring and intravenous (IV) access.

The anesthesiologist will perform a combined spinal epidural analgesia per routine with the subject in the sitting position using sterile technique at the L3-4 interspace (± one vertebral interspace). The epidural space will be found using loss of resistance technique with either 3 mL of air or saline and a 17G Touhy needle. After the epidural space is identified, the dura will be punctured with a 27G Pencan and 2.5mg of plain bupivacaine + 15 μg fentanyl will be injected. The epidural catheter will be inserted to 3-5cm into the epidural space and a test dose of 3 mL of 1.5% lidocaine + 1:200,000 epinephrine will be injected. The epidural catheter will be secured and the PCEA initiated with the standard infusion rate and patient administered boluses using 0.06% bupivacaine + 2mcg/mL fentanyl. Post-procedure vital signs will be monitored in the usual fashion.

Patients randomized to the control group will have a Foley catheter placed after the CSE is performed as is the usual practice at this institution. Their bladder volume will be assessed via ultrasonography before Foley catheter placement. The volume of urine collected in the Foley bag will be used to validate our ultrasonographic measurements.

Patients randomized to the spontaneous micturition algorithm will be assessed for spontaneous micturition and post void residual (PVR) volumes via ultrasonography at regular time intervals. First, the patient's bladder volume is measured via ultrasonography; this is followed by an attempt at spontaneous micturition. The patient will have an attempt at spontaneous micturition only if their bladder contains >100mL of urine. This ensures inability to micturate is not due to insufficient urine in the bladder prior to their attempt. An ultrasonographic measurement of their postvoid residual volume will follow their attempt to spontaneously micturate, to ensure the patient does not have urinary retention necessitating Foley catheter placement.

The first attempt at spontaneous micturition is two hours after the spinal analgesic dose is injected. A study by Campbell et al. demonstrated no urinary retention with this intrathecal dose, but it is a possibility that the spinal dose may still be present and have a differing effect than the epidural analgesic dose. As a result of this possibility, we decided that if a patient has urinary retention at this first attempt, 2 hours post injection of the spinal dose, they will have a straight catheterization and be given another chance at spontaneous micturition more than 3 hours after the spinal dose was injected. This ensures the spinal dose has completely worn off and the epidural analgesic dose is in effect before committing the patient to a bed pan or Foley catheter.

Most patients will be evaluated at least twice for ability to spontaneously micturate and have their PVR volumes accessed via ultrasonography before being assigned to either a bed pan every 2 hours or a Foley catheter placement. If the patient is able to spontaneously micturate twice and their PVR is <100mL, they will be assigned to a bed pan every 2 hours. If a patient is unable to micturate with a PVR >100mL, they will receive a Foley catheter.

The spontaneous micturition algorithm allows for a maximum of 3 attempts at micturition before a patient is committed to either a bed pan every 2 hours or Foley catheter placement. In the event that a patient is able to spontaneously micturate but has incomplete bladder emptying with a PVR 100-250mL, they will be allowed to continue in the algorithm for a third and final attempt at spontaneous micturition. If the patient is able to spontaneously micturate at this last attempt with a PVR volume <100mL, they will be assigned to a bed pan every 2 hours but if their PVR remains >100mL they will have a Foley catheter placed.

On occasion, patients need a rescue bolus of higher concentration local anesthetic during labor for breakthrough pain. If this occurs, the usual rebolus dose of up to 15mL of bupivacaine 0.125% will be given in incremental doses titrated to patient comfort. Following this rebolus, the infusion rate will be increased to 20ml/hr as is the usual practice. If a patient who was previously assigned to use a bed pan every 2 hours requires a rescue bolus of local anesthetic, their ability to spontaneously micturate will be reassessed 2 hours following the rebolus to evaluate for need for reassignment to Foley catheter placement with the higher doses of bupivacaine.

If a patient who was assigned to use a bed pan every 2 hours requires a second rebolus, they will receive another rebolus dose of up to 15mL of bupivacaine 0.125%, the concentration of the epidural bupivacaine infusion will be increased to bupivacaine 0.11% + fentanyl 2mcg/mL as is our usual practice and they will automatically be assigned to a Foley catheter placement.

If a study patient requires a cesarean delivery, a Foley catheter will be inserted at time of decision for cesarean delivery and removed 24 hours post procedure as is the standard practice at our institution.

The primary outcome (rate of positive urine culture) of this study will be assessed by collecting a twenty-four to forty-eight hour midstream urine sample and performing a urine culture. The clinical and laboratory criteria used to define a urinary tract infection in a woman immediately postpartum is unknown. If the patient is considered uncomplicated (normal female urinary physiology) then she would be treated only if she has symptoms. If the patient is considered complicated (pregnant urinary physiology) then she would be treated for bacterial growth on urine culture even if asymptomatic. For this reason and for the purpose of this study, if the patient is asymptomatic for urinary tract infection but has a positive urine culture with 50,000 colony-forming units (CFU)/mL of bacteria, the patient's obstetrician will be notified and they will likely be treated with antibiotics for suspected urinary tract infection. This is more conservative than the current guidelines for asymptomatic bacteriuria in pregnancy. If a positive urine culture is identified and patients is symptomatic (at least1 sign/symptom) with the number of colonies of bacteria exceed 10,000 CFU/ml, the obstetrician will be notified and they may be treated with antibiotics for suspected urinary tract infection. This is more conservative than the guidelines for catheter-related infections.

In addition to the primary outcome data, the following information will be collected after delivery: satisfaction with bladder treatment protocol (100 mm scale, 0 mm = not satisfied at all, 100 mm = very satisfied), total labor duration, length of stage 2, mode of delivery, presence and degree of lacerations, fetal weight, duration of Foley catheterization, time to first spontaneous void following delivery or Foley catheter removal, total fluids administered during labor and total dose of epidural analgesics.

In addition, a postvoid residual (PVR) will be assess via ultrasound at 8-24 hours following delivery or foley catheter removal to assess for postpartum urinary retention. If the PVR is found to be >100mL postpartum, this will be considered urinary retention and the obstetrician and co-investigator (urogynecologist) will be notified.

The following demographic data will also be collected: maternal age, height, weight, pre-pregnancy weight, and gestational age.

One telephone follow-up evaluation 8 weeks after delivery, the patient will be assessed for treatment of urinary tract infection and urinary retention during or after discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Term (≥37 week gestation)
* Healthy
* ASA class 1-2
* Who are being induced for labor who request labor analgesia and who successfully receive standard combined spinal epidural analgesia (verbal rating score for pain ≤ 1 after 10 min)

Exclusion Criteria:

* Women with ASA 3 or greater
* BMI ≥40 kg/m2
* Prior history of urge or stress incontinence or urinary retention before pregnancy
* Women with a history of nephrolithiasis
* Chronic urinary tract infections
* Women whose post-void residual volume as assessed by ultrasonography is found to be >100ml before epidural placement will be excluded.
* Women with an absolute or relative contraindication to the usual combined spinal epidural technique
* Failed analgesia will be excluded
* Women for whom the anesthesiologist selects an analgesic technique other than combined spinal epidural technique or fail to obtain CSF for CSE will be excluded
* Women with fetal heart rate decelerations before request for analgesia will be excluded due to increased risk of cesarean delivery.
* Women who experience inadequate labor analgesia due to nonfunctioning epidural catheter necessitating epidural replacement will be included but noted as a protocol violation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-03-22 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Bauchat, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Foley Catheter | No Foley Catheter
Started | 28 | 28
Completed | 20 | 18
Not Completed | 8 | 10
Not completed — Physician Decision | 2 | 1
Not completed — Cesarean Section | 6 | 7
Not completed — Subject withdrawal | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Foley Catheter | No Foley Catheter | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (6.8) | 33 (3.8) | 33.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Urine Culture
Description: This study will be assessed by collecting a twenty-four to forty-eight hour midstream urine sample and performing a urine culture. The clinical and laboratory criteria used to define a urinary tract infection.
Time Frame: 48 Hours
Measure: Number; unit: participants with positive urine culture
Arm/Group | Foley Catheter | No Foley Catheter
Number analyzed (Participants) | 20 | 18
participants with positive urine culture | 3 | 1
Statistical Analysis 1: Comparison: Foley Catheter vs No Foley Catheter; Test type: Superiority; p = .05, Fisher Exact — Calculated

ADVERSE EVENTS:
Time Frame: 1 day
Description: Urinary retention
Arm/Group | Foley Catheter | No Foley Catheter
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 6/20 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foley Catheter (N=20) | No Foley Catheter (N=18)
Urinary Retention (Renal and urinary disorders) | 6 (6) | 6 (6) — Urinary retention

LIMITATIONS AND CAVEATS:
The study was terminated early because of difficulty using the ultrasound device to estimate urinary bladder capacity and residual levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No